CLINICAL TRIAL: NCT02904759
Title: A Randomised, Double-blind, Placebo-controlled, Multi-centre Trial Investigating the Efficacy and Safety of Desmopressin (FE 992026) Orally Disintegrating Tablets During 12 Weeks of Treatment for Nocturia Due to Nocturnal Polyuria in Japanese Male Subjects
Brief Title: Trial of Desmopressin Orally Disintegrating Tablets (ODT) for Nocturia Due to Nocturnal Polyuria in Japanese Male Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000130
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desmopressin 25 µg (Experimental): Desmopressin ODT
  Interventions: Drug: Desmopressin
- Desmopressin 50 µg (Experimental): Desmopressin ODT
  Interventions: Drug: Desmopressin
- Placebo (Placebo Comparator): Placebo ODT
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin
  Other Names: FE 992026
  Arms: Desmopressin 25 µg; Desmopressin 50 µg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this trial is to demonstrate efficacy of desmopressin ODT against placebo for the treatment of male subjects with nocturia due to nocturnal polyuria, during 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to performance of any trial-related activity
* Man ≥20 years of age
* Nocturia symptoms present for ≥6 months prior to trial entry at Visit 1
* ≥2 nocturnal voids at the end of screening period prior to Visit 2
* Nocturnal polyuria at the end of screening period prior to Visit 2
* Bothered by nocturia on the Hsu 5-point Likert bother scale at Visit 1 and Visit 2
* Has given agreement about contraception during the trial

Exclusion Criteria:

* Evidence of any significant voiding dysfunction resulting in abnormally low bladder capacity at the end of the screening period prior to Visit 2
* History or evidence of significant obstructive sleep apnoea
* History or diagnosis of any of the following urological diseases at Visit 1:

  * Interstitial cystitis or bladder pain disorder
  * Suspicion of moderate or severe benign prostate hyperplasia (BPH), defined as international prostate symptom score (IPSS) ≥8 points and:

    * Urinary flow <5 mL/s or
    * Post-void residual volume >150 mL
  * Stress urinary incontinence or mixed incontinence, where stress incontinence is the predominant component based on prior history
  * Chronic pelvic pain syndrome
* Surgical treatment, including transurethral resection, for bladder outlet obstruction (BOO) or BPH within the past 6 months prior to Visit 1
* Symptoms of severe over-active bladder (OAB):

  * Defined as an over-active bladder symptom score (OABSS) ≥12 at Visit 1
  * Defined as a mean of >8 voids and a mean of ≥1 urgency episode per 24 hours at the end of the screening period prior to Visit 2
* Genito-urinary tract pathology that can in the investigator's opinion be responsible for urgency or urinary incontinence at Visit 1
* Complication of cancer or a history of cancer which has not been in remission for the last 5 years at Visit 1
* Current or a history of urologic malignancies, any lower urinary tract surgery, previous pelvic irradiation, or neoplasia at Visit 1
* History of any neurological disease affecting bladder function or muscle strength at Visit 1
* Habitual or psychogenic polydipsia based on medical history at Visit 1 or 24 hour urine output of >2.8 L based on the voiding diary at Visit 2
* Central or nephrogenic diabetes insipidus at Visit 1
* Syndrome of inappropriate antidiuretic hormone secretion at Visit 1
* Suspicion or evidence of cardiac failure at Visit 1
* Uncontrolled hypertension at Visit 1
* Uncontrolled diabetes mellitus at Visit 1
* Hyponatraemia (serum sodium level <135 mmol/L) at Visit 1
* Renal insufficiency at Visit 1
* Hepatic and/or biliary diseases at Visit 1
* Known or suspected hypersensitivity to desmopressin ODTs or previous desmopressin treatment for nocturia at Visit 1
* Known alcohol or substance abuse at Visit 1
* Work or lifestyle that may interfere with regular night-time sleep at Visit 1, e.g., shift workers
* Any other medical condition, laboratory abnormality, psychiatric condition, mental incapacity, or language barrier that, in the judgment of the investigator, would impair participation in the trial at Visit 1
* Use of any prohibited therapy during the trial period

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of nocturnal voids during 12 weeks of treatment | Week 1, 4, 8 and 12
  Assessed by the 3-day voiding diary

SECONDARY OUTCOMES:
Change from baseline in mean time to first awakening to void | Week 1, 4, 8 and 12
  Assessed by the 3-day voiding diary
Change from baseline in mean nocturnal urine volume | Week 1, 4, 8 and 12
  Assessed by the 3-day voiding diary
Change from baseline in mean Nocturnal Polyuria Index (NPI) | Week 1, 4, 8 and 12
  Assessed by the 3-day voiding diary
Change from baseline in Nocturia-Specific Quality-of-Life Questionnaire (N-QoL) | Week 8 and 12
Change from baseline in Insomnia Severity Index (ISI) | Week 8 and 12
Change from baseline in bother score | Week 8 and 12
  Assessed by the Hsu 5-point Likert bother scale
Frequency and severity of adverse events | From screening to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Investigational site (there may be other sites in this country), Tokyo, Japan

REFERENCES:
- [Result] Yamaguchi O, Juul KV, Falahati A, Yoshimura T, Imura F, Kitamura M. Efficacy and safety of 25 and 50 mug desmopressin orally disintegrating tablets in Japanese patients with nocturia due to nocturnal polyuria: Results from two phase 3 studies of a multicenter randomized double-blind placebo-controlled parallel-group development program. Low Urin Tract Symptoms. 2020 Jan;12(1):8-19. doi: 10.1111/luts.12276. Epub 2019 Aug 9. PMID 31397969